

#### ClinicalTrials.gov Protocol Registration and Results System (PRS) Receipt

Release Date: March 5, 2019

ClinicalTrials.gov ID: NCT03390166

# **Study Identification**

Unique Protocol ID: Tri Fluvac Vaccine phase 2/3

Brief Title: Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated

Influenza Vaccine in Healthy Thai Adults

Official Title: A Phase II/III Double Blinded, Randomized, Controlled, Non-inferiority Trial to

Evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine, in Healthy Thai Subjects Aged 18-49

Years

Secondary IDs:

# **Study Status**

Record Verification: March 2019

Overall Status: Completed

Study Start: July 24, 2017 [Actual]

Primary Completion: March 31, 2018 [Actual]

Study Completion: February 12, 2019 [Actual]

#### Sponsor/Collaborators

Sponsor: Mahidol University

Responsible Party: Principal Investigator

Investigator: Punnee Pitisuttithum [ppitisuthitham]

Official Title: Prof.

Affiliation: Mahidol University

Collaborators: The Government Pharmaceutical Organization

World Health Organization

#### Oversight

U.S. FDA-regulated Drug: No

U.S. FDA-regulated Device: No

U.S. FDA IND/IDE: No

Human Subjects Review: Board Status: Approved

Approval Number: MUTM 2017-020-01

Board Name: Ethics Comittee of the Faculty of Tropical Medicine Board Affiliation: Faculty of Tropical Medicine, Mahidol University

Phone: (662) 3069100

Email: pornpimon.ada@mahidol.ac.th

Address:

Faculty of Tropical Medicine, Mahidol University 420/6 Rajvithi road, Ratchathewi, Bangkok 10400

Thailand

Data Monitoring: Yes

FDA Regulated Intervention: No

# **Study Description**

Brief Summary: The study is aim to evaluate the immunogenicity and safety with two groups of

participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza

vaccine

Detailed Description: This is a phase II/III, non-inferiority double-blinded, randomized, controlled trial

of immunogenicity and safety with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B)

or an active comparator (licensed influenza vaccine).

A total of about 945 healthy Thai male and female adult volunteers 18 through 49 years of age; 630 participants will be randomized to receive the GPO Tri Fluvac and 315 will receive an active comparator (a 2:1 ratio) (inclusion of ~7%)

lost to follow-up).

Safety will be assessed for all participants through Day 90 after vaccination. Immunogenicity will be assessed in serum samples obtained at baseline and 21 days after vaccination in a subset of at least 586 individuals randomized to

study vaccine and 293 active comparator vaccine recipients.

#### Conditions

Conditions: Influenza

Keywords: GPO Tri Fluvac Vaccine

Tri Fluvac vaccine

# **Study Design**

Study Type: Interventional

Primary Purpose: Prevention

Study Phase: Phase 2/Phase 3

Interventional Study Model: Parallel Assignment

non-inferiority double-blinded, randomized, controlled trial

Number of Arms: 2

Masking: Double (Participant, Investigator)

double blinded

Allocation: Randomized Enrollment: 945 [Actual]

#### **Arms and Interventions**

| Arms | Assigned Interventions |
|---|---|
| Active Comparator: GPO Tri Fluvac vaccine | Biological/Vaccine: GPO Tri Fluvac vaccine |
| 630 volunteers will receive a single dose of the seasonal trivalent inactivated influenza vaccine (consisting of A/Michigan/45/2015 (H1N1)pdm-09-like virus, A/Hong Kong/4801/2014 (H3N2)-like virus, and B/Brisbane/60/2008-like virus) produced by GPO Thailand. To be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm. | The vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm. |
| Active Comparator: Licensed Influenza vaccine 315 volunteers will receive acLicensed Influenza vaccine (seasonal trivalent inactivated split virion influenza vaccine recommended for Southern Hemisphere in 2017 (consisting of A/ Michigan/45/2015 (H1N1)pdm-09-like virus, A/ Hong Kong/4801/2014 (H3N2)-like virus, and B/ Brisbane/60/2008-like virus) 0.5 mL administered intramuscularly (IM) in the deltoid muscle of the non- dominant arm. | Biological/Vaccine: Licensed influenza vaccine The comparator licensed influenza vaccine will be administered via the intramuscular route; the preferred injection site will be the deltoid of the non-dominant arm. |

#### **Outcome Measures**

Primary Outcome Measure:

1. Primary Immunogenicity Endpoint: Immune responses to the GPO Tri Fluvac and active comparator vaccine at 21 days post-injection.

null [Time Frame: 21 days post-injection]

2. Primary Safety Endpoints: Number of subjects with all Adverse Events during the study period and % of subjects with all Adverse Events during the study period

null [Time Frame: upto 90 days]

# **Eligibility**

Minimum Age: 18 Years Maximum Age: 49 Years

Sex: All

Gender Based:

Accepts Healthy Volunteers: Yes

Criteria: Inclusion Criteria:

- Age 18-49 years old on the day of screening, having Thai ID card or equivalent
- · Able to read and write in Thai and sign written informed consent form
- Able to attend all scheduled visits and to comply with all trial procedures.
- Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable, under control or unchanged for the past three months. If medication is used to treat the condition, the medication dose must have been stable for at least one month preceding vaccination.
- For female participants:

- Not breast feeding, non-pregnant (based on negative urine pregnancy test) and no plan to become pregnant up to Day 60.
- Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than one year must be willing to use effective contraceptive method to prevent pregnancy until Day 60 after vaccination. Effective methods include intrauterine device, hormonal contraceptives (oral, injectable, patch, implant, ring) or double barrier contraceptives (condom or diaphragm with spermicide). Women with credible history of abstinence may be enrolled at the discretion of the investigator

#### **Exclusion Criteria:**

- Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
- Hypersensitivity after previous administration of any vaccine.
- Having a history of H1N1, H3N2 or Flu B infection within 3 months preceding enrollment to the trial
- Vaccination against influenza in the past 6 months preceding enrollment to the trial
- Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 21 visit.
- · History of bronchial asthma, chronic lung diseases, chronic rhinitis
- · History of immunodeficiency state
- History of immunosuppression < 6 months prior to immunization</li>
- History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. gentamicin or thimerosal)
- · History of Guillain-Barré Syndrome.
- Having acute infection with fever > 38 degree Celsius or noninfectious diseases (within 72 hours) preceding enrollment in the trial
- Volunteers who have been taking immunoglobulin products or have had a blood transfusion during past 3 months before the beginning of the trial or planned receipt of such products prior to the Day 21 visit.
- Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
- Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled, or could interfere with the evaluation of the vaccine

#### Contacts/Locations

Central Contact Person: Punnee Pitisuttithum, Prof.

Telephone: (662) 6435599

Email: punnee.pit@mahidol.ac.th

Central Contact Backup:

Study Officials: Punnee Pitisuttithum, Prof.

Study Principal Investigator

Mahidol University

Locations: Thailand

Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University

Bangkok, Thailand, 10400

Contact: Punnee Pitisuttithum (662)6435599 punnee.pit@mahidol.ac.th

Principal Investigator: Punnee Pitisuttithum

Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University,

Bangkok, Thailand, 10400

Contact: Punnee Pitisuttithum 662-6445599 punnee.pit@mahidol.ac.th

Contact: 662-3549178

Principal Investigator: Punnee Pitisuttithum

# **IPDSharing**

Plan to Share IPD: Undecided

#### References

Citations:

Links:

Available IPD/Information:

U.S. National Library of Medicine | U.S. National Institutes of Health | U.S. Department of Health & Human Services

### Statistical Analysis Plan (SAP)

#### For

#### Government Pharmaceutical Organization (GPO)

A Phase II/III Double Blinded, Randomized, Controlled, Non-inferiority Trial to Evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated Split Virion Influenza Vaccine, in Healthy THAI Subjects Aged 18-49 years.

### Prepare by

Montida Auayporn, Statistician, BIOPHICS

Center of Excellence for Biomedical and Public Health Informatics (BIOPHICS)

Faculty of Tropical Medicine, Mahidol University

Rajavithi Campus, Bangkok 10400

Version 1.0, 12 February 2018

| Study Title: | A Phase II/III Double Blinded, Randomized, Controlled, Non-inferiority trial to evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated split virion Influenza vaccine, in healthy THAI subjects aged 18 - 49 years. |
|---|---|
| Study Protocol: | GPO Tri Fluvac Vaccine (Phase II/ III) |
| SAP Approval<br>Date: | 12 FEB 2018 |
| SAP Version # and Date: | Version 1.0, 12 February 2018 |

| SIGN | VA | TI | R | ES |
|------|------|----|---|----|
| | 72 A | | | |

SUBMITTED BY: I have authored this document and submit it for approval.

| Montida A. | DATE:_ | 12 FEB 2018 |
|---|---|---|
| Montida Auayporn | | |
| Statistician | | |
| BIOPHICS | | |
| Center of Excellence for Biomedical and Public Health | Informatics | |

REVIEWED BY: I have reviewed this document and find it to be accurate and acceptable.

My Cent

DATE: 12 FEB 2018

Saranath Lawpoolsri

**Chief of Biomedical Informatics** 

**BIOPHICS** 

Center of Excellence for Biomedical and Public Health Informatics

# **Table of Contents**

| Study Synopsis |
|---|
| Study Summary |
| FREF 01: Study Profile |
| FREF 02: Number and Percentage of Cases with Adverse Events |
| FREF 03: Number and Percentage of Adverse Events by Systemic Organ Class (by Each Group) |
| FREF 04: Number and Percentage of Cases with Adverse Events by Systemic Organ Class (by Each |
| Group) |
| FREF 05: Summary Number and Percentage of Cases by Temperature Grading and Follow up Visit 10 |
| FREF 06: Summary Number and Percentage of Cases by Temperature Grading at Post Immunization |
| FREF 07: Number and Percentage of Local Reaction Grading at Post Immunization |
| FREF 08: Number and Percentage of Systemic Reaction Grading at Post Immunization |
| TREF 01: Summary of Seroconversion, Seroprotection, GMT and GMFRs |
| TREF 02: Summary of Non-inferiority Established Based on Seroconversion Rate Differences and GMT Ratios |
| TREF 03: Summary Immunogenicity Result: GMT Ratio |
| TREF 04: Summary Immunogenicity Result: Seroconversion Rate (SCR) Difference |
| FREF 09: Summary Geometric Mean Titer (GMT) with 95% CI Against Each of Three Vaccine 1 |
| Antigens at Day 211 |
| FREF 10: Summary Geometric Mean Titer (GMT) with 95% CI Against Each of Three Vaccine 1 |
| Antigens at Day 901 |
| FREF 11: Summary Percentage of Seroprotection with 95% CI Against Each of Three Vaccine 13 |
| Antigens at Day 2113 |
| FREF 12: Summary Percentage of Seroprotection with 95% CI Against Each of Three Vaccine 13 |
| Antigens at Day 901 |
| FREF 13: Summary Percentage of Seroconversion with 95% CI Against Each of Three Vaccine Antigens at Day 21 |
| FREF 14: Summary Percentage of Seroconversion with 95% CI Against Each of Three Vaccine 19 |
| Antigens at Day 9019 |
| FREF 15: Summary Non-Inferiority Trial of GMTs Ratio and 95% Confidence Interval at Day 21 20 |
| FREF 16: Summary Non-Inferiority Trial of GMTs Ratio and 95% Confidence Interval at Day 21 at Day 90 |
| FREF 17: Summary Non-Inferiority Trial of Seroconversion Difference (%) and 95% Confidence Interval at Day 21 |

| | FREF 18: Summary Non-Inferiority Trial of Seroconversion Difference (%) and 95% Confidence Interval at Day 90 | 23 |
|---|---|---|
| 1. | General Subject Characteristics at Screening | 24 |
| | TREF 1.1: Demographics and Subject Characteristics at Screening by GPO Tri fluvac and Active Comparator Group | 25 |
| | TREF 1.2: Medical History at Screening by GPO Tri fluvac and Active Comparator Group | 26 |
| | TREF 1.3: Vital Sign at Screening by GPO Tri fluvac and Active Comparator Group | 27 |
| | TREF 1.4: Physical Examination at Screening by GPO Tri fluvac and Active Comparator Group | 29 |
| | TREF 1.5: Urine Pregnancy Test at Prior Immunization (Day 0) | 30 |
| 2. | Safety Assessment | 31 |
| | TREF 2.1: Summary of Treatment Emergent Adverse Events by GPO Tri fluvac and Active Comparator Group | 32 |
| | TREF 2.2: Comparison of Maximum Severity Grade of Adverse Event by GPO Tri fluvac and Active Comparator Group | |
| | TREF 2.3: Summary of Adverse Events Classified by MedDRA term | 34 |
| | TREF 2.4: Summary of Adverse Events Related to Treatment | 34 |
| | TREF 2.5: Summary of Adverse Events with Definitely Related and / or Severe | 35 |
| | TREF 2.6: Summary Number of Subjects with Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group | 36 |
| | TREF 2.7: Vital Sign of Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Grou | • |
| | TREF 2.8: Physical Examination of Illness like Influenza (ILI) Events by GPO Tri fluvac and Activ Comparator Group | ⁄e |
| 3. | Post Immunization Reaction | 41 |
| | TREF 3.1: Comparison of Temperature Grading at Follow up Visit by GPO Tri Fluvac and Active Comparator Group | 42 |
| | TREF 3.2: Comparison of Temperature Grading at Post Immunization by GPO Tri Fluvac and Active Comparator Group | |
| | TREF 3.3: Vital Sign at Follow up Visit by GPO Tri Fluvac and Active Comparator Group | 44 |
| | TREF 3.4: Physical Examination by GPO Tri Fluvac and Active Comparator Group | 46 |
| | TREF 3.5: Comparison of Maximum Grade of Any Local Reaction at Post Immunization by GPO T fluvac and Active Comparator Group | |
| | TREF 3.6: Comparison of Local Reaction at Post Immunization each Follow up Time by GPO Tri Fluvac and Active Comparator Group | 49 |
| | TREF 3.7: Comparison of Maximum Grade of Local Reaction by Symptom at Post Immunization b<br>GPO Tri fluvac and Active Comparator Group | - |

| | TREF 3.8: Comparison Number of Subject by Number of Local Reaction Days at Post Immunization GPO Tri fluvac and Active Comparator Group |
|---|---|
| | TREF 3.9: Comparison Number of Subjects by Number of Local Reaction at Post Immunization GPO Tri fluvac and Active Comparator Group |
| | TREF 3.10: Comparison of Maximum Grade of Any Systemic Reaction at Post Immunization by GPO Tri fluvac and Active Comparator Group |
| | TREF 3.11: Comparison of Systemic Reaction at Post Immunization each Follow up Time by GPO Tri fluvac and Active Comparator Group |
| | TREF 3.12: Comparison of Maximum Grade of Systemic Reaction by Symptom at Post Immunization by GPO Tri fluvac and Active Comparator Group |
| | TREF 3.13: Comparison Number of Subject by Number of Systemic Reaction Days at Post Immunization GPO Tri fluvac and Active Comparator Group |
| | TREF 3.14: Comparison Number of Subjects by Number of Systemic Reaction at Post Immunization between GPO Tri fluvac and Active Comparator Group |
| 4. | Immunogenicity 60 |
| | TREF 4.1: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90 |
| | TREF 4.2: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator at Any Day |
| | TREF 4.3: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer < 1:10 |
| | TREF 4.4: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer $\geq 1:10$ |
| | TREF 4.5: Comparing Seroprotective Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90 |
| | TREF 4.6: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer < 1:10 |
| | TREF 4.7: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer $\geq 1:10$ |
| | TREF 4.8: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group |
| | TREF 4.9: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer < 1:10 |
| | TREF 4.10: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer $\geq 1:10$ |
| | TREF 4.11: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group |

| • | Rs) of Immune Response by GPO Tri fluvac and ccination HI Antibody Titer < 1:10 | 72 |
|---|---|---|
| ` | Rs) of Immune Response by GPO Tri fluvac and ccination HI Antibody Titer $\geq 1:10$ | 73 |
| 5. Concomitant Medication | | 74 |
| • | According to WHO DD by GPO Tri fluvac and Activ | |
| APPENDICES | | 76 |
| Appendix 01: Listing of Subjects were Excluded | l from Analysis | 76 |
| Appendix 02: Listing of Past Medical History ar | nd Pre-existing Condition in Last 6 Months | 76 |
| Appendix 03: Listing of Past Immunization Hist | ory in Last 6 Months | 76 |
| Appendix 04: Listing of Local Reaction at Post | Immunization | 77 |
| Appendix 05: Listing of Systemic Reaction at Po | ost Immunization | 77 |
| Appendix 06: Listing of Adverse Event | | 78 |
| Appendix 07: Listing of Illness like Influenza (I | LI) | 78 |
| Appendix 08: Listing of Concomitant Medicatio | n | 79 |
| Appendix 09: List of HAI Assay (Flu A H1 Ant | igen) | 80 |
| Appendix 10: List of HAI Assay (Flu A H3 Anti | igen) | 80 |

#### **Study Synopsis**

**Title:** A Phase II/III Double Blinded, Randomized, Controlled, Non-inferiority trial to evaluate the Immunogenicity and Safety of Tri Fluvac, a Seasonal Trivalent Inactivated split virion Influenza vaccine, in healthy Thai subjects aged 18 – 49 years.

Protocol #: GPO Tri Fluvac Vaccine Phase II/III

#### **Description of Study Design:**

This is a phase II/III, non-inferiority double-blinded, randomized, controlled trial of immunogenicity, safety and preliminary efficacy with two groups of participants who will received a seasonal trivalent split, inactivated influenza vaccine (A/H1N1; A/H3N2 and B) or an active comparator (licensed influenza vaccine).

A total of about 945 healthy Thai male and female adult volunteers 18 through 49 years of age; 630 participants will be randomized to receive vaccine and 315 will receive an active comparator (a 2:1 ratio) (inclusion of  $\sim$ 7% lost to follow-up).

Safety will be assessed for all participants through Day 90 after vaccination. Immunogenicity will be assessed in serum samples obtained at baseline and 21 days after vaccination in a subset of at least 630 individuals randomized to study vaccine and 315 active comparator vaccine recipients.

#### Study Hypothesis:

Immunogenicity: A single dose of the GPO seasonal trivalent split, inactivated influenza vaccine will induce immune responses measured by HI assay to each of the three vaccine antigens and will be non-inferior to active licensed comparator vaccine.

Safety: A single dose of the GPO seasonal trivalent split, inactivated influenza vaccine will be safe and well tolerated in adults 18 to 49 years of age.

**Study Objectives:** 

Primary objective

#### Immunogenicity:

To evaluate the immunological non-inferiority seroconversion rate (using HI assay) and Geometric Mean Titre (GMT) of the GPO seasonal trivalent split, inactivated influenza vaccine compared to active comparator vaccine for each of the three vaccine antigens, three weeks after immunization (Day 21) and at the end of follow up period (Day 90).

#### Safety:

To evaluate the safety profile of a single intramuscular dose of the GPO seasonal trivalent split, inactivated influenza vaccine in adults 18 to 49 years of age. To compare the solicited symptoms, AE and

SAE between subjects who will receive GPO trivalent split, inactivated influenza vaccine and those who will receive active comparator vaccine.

#### Secondary objective

To evaluate the HI responses at 3 weeks after immunization in participants with or without preexisting HI antibody.

# Study Endpoints and Statistical Analysis:

#### **Primary Immunogenicity Endpoint:**

Immune responses to the GPO Tri Fluvac and active comparator vaccine at 21 days post-injection will be analyzed by the following:

- Number and percentage of participants with seroconversion against each of the three vaccine antigens. Seroconversion is defined as a serum HI antibody titer meeting the following four fold rising criteria:
  - Pre-vaccination titer <1:10 and a post-vaccination titer measured on Day21 of ≥1:40; or
  - Pre-vaccination titer ≥1:10 and at least a four-fold increase in post vaccination measured on Day 21.
- Geometric mean titers (GMTs) of serum HI antibodies pre- (Day 0) and post-vaccination (Day 21) for each of the three vaccine antigens.

Note that titers below the lowest limit of quantitation (i.e., below the starting dilution of assay reported as "< 10") will be set to half that limit (i.e., 10/2 = 5). If a titer is reported as greater or equal to the upper limit of the assay, it will be set to that limit. The analyses will be performed on the Total Vaccinated cohort (ITT) and According to Protocol (ATP) cohort for immunogenicity.

- The Total Vaccinated cohort will include all subjects with a documented vaccine administration.
- The ATP cohort for immunogenicity will include all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity outcome variables were available for antibodies against at least one study vaccine antigen component after vaccination.

#### **Primary Safety Endpoints:**

Counts and percentages of subjects with solicited local and systemic reactions during the three days post-injection. In addition, all adverse events (AE) and serious adverse events (SAEs), and new onset of chronic diseases (NOCDs) will be collected for the entire study period. Specifically, the following safety parameters will be monitored and analyzed in terms of the number and proportion of participants reporting the following events will be assessed:

- Solicited local adverse events, including redness/erythema, swelling/induration, pain and limitation of arm movement within 30 minutes of vaccination and over the 3-day period post vaccination (Day 0-3).
- Solicited systemic adverse events, including fever, fatigue/malaise, muscle aches, joint aches, chills, nausea and headache within 30 minutes of vaccination and over the 3-day period post vaccination (Day 0-3).
  - Unsolicited adverse events (AEs) occurring within 90 days post vaccination.
  - Serious Adverse Events (SAE) occurring during the entire study period (Days 0-90).

Counts of all events will be reported and summarized according to event severity, as "any local AE", or "any systemic AE", and by relationship to administration of study product, as deemed by a blinded study clinician. Percentages of participants experiencing each reaction or event, or at least one reaction or event will be calculated along with two-sided exact 95% CIs. The percentage of participants with solicited AE and SAEs will be compared between vaccine and comparator groups and a two-sided p-value of 0.05 will be considered statistically significant.

#### Inferential analyses

GMT ratios (GMT active comparator vaccine/GMT GPO TRI FLUVAC) and difference of seroconversion rate (with two-sided 95% CI) related to the comparisons of interest will be computed. Acceptance value of GMT ratios at  $\leq 1.5$  and/or difference of seroconversion rate at  $\leq 10\%$  for the upper bound of the 95% CI will be considered for non-inferiority.

#### Secondary Immunogenicity Endpoints and analysis:

The secondary immunogenicity endpoints will be analyzed by the following:

- Number and percentage of participants with a HI antibody titer ≥1:40 (seroprotective level) to each of the three vaccine antigens measured on Day 21 and Day 90.
- Number and percentage of participants who develop at least a four-fold increase in HI antibody titers to each of the vaccine antigen post-vaccination measured on Day 21 and Day 90 segregated by prevaccination HI antibody titers (<1:10 or ≥1:10).
- Geometric mean fold rises (GMFRs) of serum HI antibodies (post vaccination/ pre-vaccination) for each of the three vaccine antigens.
- GMTs of serum HI antibodies pre- (Day 0) and post-vaccination (Day 21 and Day 90) for each of the three vaccine antigens segregated by pre-vaccination HI antibody titers (<1:10 or  $\ge1:10$ ).
- GMFRs of serum HI antibodies (post-vaccination/pre-vaccination) for each of the three vaccine antigens segregated by pre-vaccination HI antibody titers (<1:10 or  $\ge1:10$ ).

#### **Study Population:**

About 945 male and female adults, 18 to 49 years of age

### Eligibility Criteria:

#### Inclusion:

- Age 18-49 years old on the day of screening, having Thai ID card or equivalent
- Able to read and write in Thai and sign written informed consent form
- Able to attend all scheduled visits and to comply with all trial procedures.
- Healthy or medically stable, as established by medical history and physical examination. For individuals with medical conditions, symptoms/signs, if present must be stable under control or unchanged for the past three months. If medication is used to treat the condition, the medication dose must have been stable for at least one month preceding vaccination.

#### For female participants:

- Not breast feeding, non-pregnant (based on negative urine pregnancy test) and no plan to become pregnant up to Day 60.
- Women who are not surgically sterile (hysterectomy or tubal ligation) or post-menopausal for more than one year must be willing to use effective contraceptive method to prevent pregnancy until Day 60 after vaccination. Effective methods include intrauterine device, hormonal contraceptives (oral, injectable, patch, implant, ring) or double barrier contraceptives (condom or diaphragm with spermicide). Women with credible history of abstinence may be enrolled at the discretion of the investigator.

#### Exclusion:

- Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
  - Hypersensitivity after previous administration of any vaccine.
- Having a history of H1N1, H3N2 or Flu B infection as H1N1, H3N2, or Flu B within 3 months preceding enrollment to the trial
  - Vaccination against influenza in the past 6 months preceding enrollment to the trial
- Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 21 visit.
  - History of bronchial asthma, chronic lung diseases, chronic rhinitis
  - History of immunodeficiency state
  - History of immunosuppression < 6 months prior to immunization
- History of anaphylactic or other allergic reactions to influenza vaccine or any vaccine component or excipient (e.g. gentamicin or thimerosal)
  - History of Guillain-Barré Syndrome.

Page 5 of 80

- Having acute infection with fever > 38 degree Celsius and noninfectious diseases (within 72

hours) preceding enrollment in the trial

- The volunteers who have been taking immunoglobulin products or have had a blood transfusion

during past 3 months before the beginning of the trial or planned receipt of such products prior to the Day

21 visit. Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial

procedures

- Any condition that in the opinion of the investigator would pose a health risk to the subject if

enrolled, or could interfere with the evaluation of the vaccine

Phase: II/III

**Study Duration:** 

Approximately 1 year

**Participation Duration:** 

About three to four months per participant

Description of Agent or Intervention:

The vaccine is a seasonal trivalent inactivated split virion influenza vaccine recommended for

Southern hemisphere in 2017 (consisting of A/Michigan/45/2015(H1N1)pdm-09-like virus, A/Hong

Kong/4801/2014 (H3N2)-like virus, and B/Brisbane/60/2008-like virus) produced by The Government

Pharmaceutical Organization (GPO), Thailand. Each dose of Tri Fluvac contains a total of 45

micrograms (µg) hemagglutinin (HA) per 0.5 ml dose (15 µg HA per strain per dose), to be administered

by intramuscular (IM) injection. Tri Fluvac is manufactured and formulated into a multiple-dose vial

vaccine (2 doses) using thimerosal at relatively low concentration as preservative (≤ 7.5 μg mercury/

dose). Each 0.5 ml dose of vaccine may contain residual amounts of ovalbumin ( $\leq 5.0 \,\mu g$ ),

formaldehyde ( $\leq 50 \mu g$ ), tween  $80 (\leq 250 \mu g)$ , triton x-100 ( $\leq 5 \mu g$ ) and gentamic (not more than 0.05

μg). The vaccine should be administered as a single 0.5ml intramuscular injection, preferably in the

region of the deltoid muscle of the upper arm.

**Description of active comparator vaccine:** 

a Licensed Influenza vaccine (seasonal trivalent inactivated split virion influenza vaccine

recommended for Southern hemisphere in 2017 (consisting of A/Michigan/45/2015 (H1N1) pdm-09-like

virus, A/Hong Kong/4801/2014 (H3N2) - like virus, and B/Brisbane/60/2008-like virus) 0.5 mL

administered intramuscularly (IM) in the deltoid muscle.

# **Study Summary**

FREF 01: Study Profile





FREF 02: Number and Percentage of Cases with Adverse Events



FREF 03: Number and Percentage of Adverse Events by Systemic Organ Class (by Each Group)



FREF 04: Number and Percentage of Cases with Adverse Events by Systemic Organ Class (by Each Group)



FREF 05: Summary Number and Percentage of Cases by Temperature Grading and Follow up Visit



FREF 06: Summary Number and Percentage of Cases by Temperature Grading at Post Immunization



FREF 07: Number and Percentage of Local Reaction Grading at Post Immunization

Note: Erythema and Induration will be not included.



FREF 08: Number and Percentage of Systemic Reaction Grading at Post Immunization

TREF 01: Summary of Sero-conversion, Sero-protection, GMT and GMFRs

| Study Group | Flu A H1 antibody titer | | |
|---|---|---|---|
| | • | Flu A H3 antibody titer | Flu B antibody titer |
| Tri fluvac (N= ) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| Comparator (N=) | xx.xx (xx.xx, xx.xx) | XX.XX (XX.XX, XX.XX) | xx.xx (xx.xx, xx.xx) |
| P –value = | X.XXXX | X.XXXX | X.XXXX |
| Tri fluvac (N= ) | | | |
| Comparator (N= ) | | | |
| P –value = | | | |
| Tri fluvac (N= ) | | | |
| Comparator (N= ) | | | |
| P –value = | | | |
| Tri fluvac (N= ) | | | |
| Comparator (N= ) | | | |
| Tri fluvac (N= | | | |
| Comparator (N= ) | | | |
| P –value = | | | |
| Tri fluvac (N= ) | | | |
| Comparator (N= ) | | | |
| P –value = | | | |
| | Comparator (N=) P-value = Tri fluvac (N=) Comparator (N=) P-value = Tri fluvac (N=) Comparator (N=) P-value = Tri fluvac (N=) Comparator (N=) Tri fluvac (N=) Comparator (N=) Tri fluvac (N=) Comparator (N=) | Comparator (N=) xx.xx (xx.xx, xx.xx) P-value = x.xxxx Tri fluvac (N=) Comparator (N=) P-value = Tri fluvac (N=) P-value = Tri fluvac (N=) Comparator (N=) Comparator (N=) Tri fluvac (N=) Comparator (N=) Tri fluvac (N=) Comparator (N=) P-value = Tri fluvac (N=) Comparator (N=) | Comparator (N= ) xx.xx (xx.xx, xx.xx) xx.xx (xx.xx, xx.xx) P -value = x.xxxx x x.xxxx Tri fluvac (N= ) Comparator (N= ) P -value = Tri fluvac (N= ) Comparator (N= ) P -value = Tri fluvac (N= ) Comparator (N= ) Tri fluvac (N= ) Comparator (N= ) P -value = Tri fluvac (N= ) Comparator (N= ) Comparator (N= ) Comparator (N= ) |

TREF 01: Summary of Sero-conversion, Sero-protection, GMT and GMFRs (Continue)

| Measure | Study Group | HAI Assay | | |
|---|---|---|---|---|
| | | Flu A H1 antibody titer | Flu A H3 antibody titer | Flu B antibody titer |
| GMT <sup>c</sup> | Tri fluvac (N= ) | | | |
| | Comparator (N= ) | | | |
| | P –value = | | | |
| GMFRs d | Tri fluvac (N= ) | | | |
| | Comparator (N= ) | | | |

Note: a Sero-conversion is defined as 4 fold rising titer from baseline (Day 0). Values are the percent of subjects in each group (with 95% CI).

b Sero-protection is defined as a HAI titer  $\geq$  40; values are the percent of subjects in each group (95% CI) with a HAI titer  $\geq$  40.

<sup>&</sup>lt;sup>c</sup> Values are the geometric means titer (GMT) (with 95% CI) for the subjects in each group.

<sup>&</sup>lt;sup>d</sup> Geometric Mean Fold Rises (GMFR) is the geometric mean of the ratios of post - vaccination to the pre-vaccination (Day 0)

<sup>-</sup> Seroconversion rate, seroprotection rate and GMTs will be compared between Tri Fluvac and comparator group.

TREF 02: Summary of Non-inferiority Established Based on Seroconversion Rate Differences and GMT Ratios

| Measure | Study Group | HAI Assay | | |
|---|---|---|---|---|
| Measure | Study Group | Flu A H1 antibody titer | Flu A H3 antibody titer | Flu B antibody titer |
| Day 0 | | | | |
| GMT <sup>c</sup> | Tri Fluvac (N= ) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Comparator (N= ) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| Day 21 | | | | |
| Seroconversion Rate <sup>a</sup> | Tri Fluvac (N= ) | XX.XX% (XX.XX%, XX.XX%) | XX.XX% (XX.XX%, XX.XX%) | xx.xx% (xx.xx%, xx.xx%) |
| | Comparator (N= ) | XX.XX% (XX.XX%, XX.XX%) | XX.XX% (XX.XX%, XX.XX%) | xx.xx% (xx.xx%, xx.xx%) |
| Difference in Seroconversion Rate <sup>b</sup> | | XX.XX% (XX.XX%, XX.XX%) | XX.XX% (XX.XX%, XX.XX%) | xx.xx% (xx.xx%, xx.xx%) |
| GMT <sup>c</sup> | Tri Fluvac (N= ) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| | Comparator (N=) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| GMT Ratio <sup>d</sup> | | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) | xx.xx (xx.xx, xx.xx) |
| Day 90 | | | | |
| Seroconversion Rate <sup>a</sup> | Tri Fluvac (N= ) | | | |
| | Comparator (N= ) | | | |
| Difference in Seroconversion Rate <sup>b</sup> | | | | |
| GMT ° | Tri Fluvac (N= ) | | | |
| | Comparator (N= ) | | | |
| GMT Ratio <sup>d</sup> | | | | |

Note: a Sero-conversion is defined as 4 fold rising titer from baseline (Day 0). Values are the percent of subjects in each group (with 95% CI).

 $<sup>^{\</sup>rm b}$  Percent difference in Seroconversion rate (with 95% CI). Clinical margin  $\leq$  10 %

<sup>&</sup>lt;sup>c</sup> Values are the geometric means titer (GMT) (with 95% CI) for the subjects in each group.

<sup>&</sup>lt;sup>d</sup> Values are the geometric means of the individual at Day 21 and Day 90 of Active comparator vaccine/ GPO Tri Fluvac HAI ratio. Clinical margin ≤ 1.5

<sup>-</sup> Non-inferiority criteria based on GMT ratio if the ratio for each HI assay at  $\leq 1.5$  and / or difference of seroconversion rate at  $\leq 10\%$  for the upper bound of the 95% CI.

TREF 03: Summary Immunogenicity Result: GMT Ratio

| Day | Antibody Titer | GMT Ratio<br>[Comparator/ Tri Fluvac]<br>(95% CI) | Non- inferiority<br>(Upper bound of the two-sided 95%<br>CI of GMT ratio ≤ 1.5) |
|---|---|---|---|
| Day 21 | Flu A H1 | x.xx(x.xx - x.xx) | Yes / No |
| | Flu A H3 | | |
| | Flu B | | |
| Day 90 | Flu A H1 | | |
| | Flu A H3 | | |
| | Flu B | | |

TREF 04: Summary Immunogenicity Result: Sero-conversion Rate (SCR) Difference

| Day | Antibody Titer | SCR (%) difference<br>[Comparator-Tri Fluvac]<br>(95% CI) | Non- inferiority<br>(Upper bound of the two-sided 95%<br>CI of SCR Difference ≤ 10%) |
|---|---|---|---|
| Day 21 | Flu A H1 | x.xx(x.xx - x.xx) | Yes / No |
| | Flu A H3 | | |
| | Flu B | | |
| Day 90 | Flu A H1 | | |
| | Flu A H3 | | |
| | Flu B | | |

**Note**: Non-inferiority criteria based on GMT ratio if the ratio for each HI assay at  $\leq 1.5$  and / or difference of seroconversion rate at  $\leq 10\%$  for the upper bound of the 95% CI.



FREF 09: Summary Geometric Mean Titer (GMT) with 95% CI Against Each of Three Vaccine
Antigens at Day 21



FREF 10: Summary Geometric Mean Titer (GMT) with 95% CI Against Each of Three Vaccine Antigens at Day 90



FREF 11: Summary Percentage of Seroprotection with 95% CI Against Each of Three Vaccine Antigens at Day 21



FREF 12: Summary Percentage of Seroprotection with 95% CI Against Each of Three Vaccine Antigens at Day 90



FREF 13: Summary Percentage of Seroconversion with 95% CI Against Each of Three Vaccine Antigens at Day 21



FREF 14: Summary Percentage of Seroconversion with 95% CI Against Each of Three Vaccine Antigens at Day 90



FREF 15: Summary Non-Inferiority Trial of GMTs Ratio and 95% Confidence Interval at Day 21  $\,$ 

-  $\Delta = \text{margin}$ 



FREF 16: Summary Non-Inferiority Trial of GMTs Ratio and 95% Confidence Interval at Day 90  $\,$ 

-  $\Delta = \text{margin}$ 



FREF 17: Summary Non-Inferiority Trial of Seroconversion Difference (%) and 95% Confidence Interval at Day 21

-  $\Delta = margin$ 



FREF 18: Summary Non-Inferiority Trial of Seroconversion Difference (%) and 95% Confidence Interval at Day 90

-  $\Delta = margin$ 

# 1. General Subject Characteristics at Screening

- TREF 1.1: Demographics and Subject Characteristics at Screening by GPO Tri fluvac and Active Comparator Group
- TREF 1.2: Medical History at Screening by GPO Tri fluvac and Active Comparator Group
- TREF 1.3: Vital Sign at Screening by GPO Tri fluvac and Active Comparator Group
- TREF 1.4: Physical Examination at Screening by GPO Tri fluvac and Active Comparator Group
- TREF 1.5: Urine Pregnancy Test at Prior Immunization (Day 0)

TREF 1.1: Demographics and Subject Characteristics at Screening by GPO Tri fluvac and Active Comparator Group

| | | Screen Failed | Enrolled | |
|---|---|---|---|---|
| | All Subjects | | Tri fluvac | Comparator |
| | (N = xx) | (N = xx) | (N = xx) | (N = xx) |
| Sex, n (%) | | | | |
| Male | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| Female | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| P- value = x.xxxx | | | | |
| Age (years), n (%) | | | | |
| n | | | | |
| Mean(SD) | | | | |
| Median | | | | |
| Min, Max | | | | |
| P- value = | | | | |
| Birth place, n (%) | | | | |
| Bangkok and | | | | |
| Other | | | | |
| P- value = | | | | |
| Level of education, n (%) | | | | |
| No education | | | | |
| Primary school | | | | |
| Secondary | | | | |
| Vocational | | | | |
| Bachelor degree | | | | |
| Higher than | | | | |
| P- value = | | | | |
| Occupation, n (%) | | | | |
| No occupation | | | | |
| Student | | | | |
| Government | | | | |
| Employee | | | | |
| Merchant | | | | |

Note: - Enrollment cases will be compared between GPO Tri fluvac and Active Comparator.

Own business

P- value =

Other
TREF 1.2: Medical History at Screening by GPO Tri fluvac and Active Comparator Group

| | | | | Enrolled | |
|---|---|---|---|---|---|
| | | All Subjects<br>(N=xx) | Screen Failed<br>(N=xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| In the last 6 months, p | ast medical hist | ory and pre-exi | sting condition, n | (%) | |
| Yes | | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| No | | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| P- value = | X.XXXX | | | | |
| In the last 6 months, p | oast immunizatio | on history, n (% | ) | | |
| Yes | | | | | |
| No | | | | | |

Note: - Enrolled cases will be compared between GPO Tri fluvac and Active Comparator.

- Past medical and immunization history will be showed as list in appendix.

TREF 1.3: Vital Sign at Screening by GPO Tri fluvac and Active Comparator Group

| | | | | Enr | olled |
|---|---|---|---|---|---|
| | | All subjects | Screen Failed | Tri fluvac | Comparator |
| | | (N = xx) | (N = xx) | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ |
| Height (cm.) | | | | | |
| n | | XX | XX | XX | XX |
| Mean(SD) | | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | | XX.XX | XX.XX | XX.XX | XX.XX |
| Min, Max | | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX | XX.XX, XX.XX |
| | P- value = $x.xxxx$ | | | | |
| Weight (kg.) | | | | | |
| n | | | | | |
| Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| <b>,</b> | P- value = | | | | |
| BMI | | | | | |
| n | | | | | |
| Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| | P- value = | | | | |
| Temperature | (°C) | | | | |
| n | , , | | | | |
| Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| 1,111, 1,141 | P- value = | | | | |
| Pulse (Beats p | | | | | |
| n | , | | | | |
| Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| wiii, wax | P- value = | | | | |
| Blood Pressur | | | | | |
| Systolic (mml | | | | | |
| | ing) | | | | |
| n<br>Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| wiii, wax | D 1 | | | | |
| | P- value = | | | | |

TREF 1.3: Vital Sign at Screening by GPO Tri fluvac and Active Comparator Group (Continue)

| | | All subjects $(N = xx)$ | Screen Failed<br>(N = xx) | Tri fluvac<br>(N = xx) | Comparator<br>(N = xx) |
|---|---|---|---|---|---|
| Diastolic | | | | | |
| n | | | | | |
| Mean(SD) | | | | | |
| Median | | | | | |
| Min, Max | | | | | |
| | P- value = | | | | |

Note: Enrolled cases will be compared between GPO Tri fluvac and Active Comparator.

TREF 1.4: Physical Examination at Screening by GPO Tri fluvac and Active Comparator Group

| | | | Enr | olled |
|---|---|---|---|---|
| | All subjects (N=xx) | Screen Failed<br>(N=xx) | Tri fluvac<br>(N = xx) | Comparator $(N = xx)$ |
| HEENT, n (%) | | | | |
| Normal | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| Abnormal | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| P- value = $x.xxxx$ | | | | |
| Lungs, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Cardiovascular, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Gastrointestinal, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Musculoskeletal, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Skin, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Neurologic, n (%) | | | | |
| Normal | | | | |
| Abnormal | | | | |
| P- value = | | | | |
| Other | | | | |
| Normal | | | | |
| Abnormal | | | | |
| p-value = | | | | |

Note: - Enrolled cases will be compared between GPO Tri fluvac and Active Comparator.

TREF 1.5: Urine Pregnancy Test at Prior Immunization (Day 0)

| | Enr | olled |
|-----------------------------|----------------------|----------------------|
| | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
| Urine Pregnancy Test, n (%) | | |
| Positive | | |
| Negative | | |
| P- value | = | |

Note: - Enrolled cases will be compared between GPO Tri fluvac and Active Comparator.

- A urine pregnancy test will be done in females on Day 0 prior to vaccination.

# 2. Safety Assessment

#### Adverse Event

- TREF 2.1.: Summary of Treatment Emergent Adverse Event by GPO Tri fluvac and Active Comparator Group
- TREF 2.2: Comparison of Maximum Severity Grade of Adverse Event by GPO Tri fluvac and Active Comparator Group
- TREF 2.3: Summary of Adverse Events Classified by MedDRA term
- TREF 2.4: Summary of Adverse Events Suspected to be Related to Treatment
- TREF 2.5: Summary of Adverse Events with Definitely Related and / or Severe

## Illness like Influenza (ILI)

- TREF 2.6: Summary Number of Subjects with Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group
- TREF 2.7: Vital Sign of Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group
- TREF 2.8: Physical Examination of Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group
- TREF 2.9: Summary RT- PCR Test for Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group

TREF 2.1: Summary of Treatment Emergent Adverse Events by GPO Tri fluvac and Active Comparator Group

| | EV | EVENT | | ASE |
|---|---|---|---|---|
| | Tri fluvac<br>(N = xx) | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| Experienced AE, n (%) | | | | |
| • AE suspected to be not related to Treatment | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |
| • AE **suspected to be related to Treatment | | | | |
| Experienced SAE, n (%) | | | | |
| • SAE suspected to be not related to Treatment | | | | |
| SAE **suspected to be related to Treatment | | | | |

Note: - Percentage of events will be calculated from all events of AE.

- Percentage of cases will be calculated from all cases.
- \*\* suspected to be related treatment = Probably not related ,Probably related, Definitely related

TREF 2.2: Comparison of Maximum Severity Grade of Adverse Event by GPO Tri fluvac and Active Comparator Group

| Severity | Tri fluvac<br>(N = xx)<br>n (%) | Comparator<br>(N = xx)<br>n (%) |
|---|---|---|
| Mild | xx(xx.xx) | xx(xx.xx) |
| Moderate | | |
| Severe | | |
| Life-threatening | | |
| P- value = $x.xxxx$ | | |

Note: Summary by case who had any AEs

TREF 2.3: Summary of Adverse Events Classified by MedDRA term

| | Event | | Event | Case | |
|---|---|---|---|---|---|
| System Organ Class Term (SOC) | Preferred Term(PT) | Tri fluvac<br>(N = xx) | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| | | n (%) | n (%) | n (%) | n (%) |
| | | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |

TREF 2.4: Summary of Adverse Events Related to Treatment

| | | Event | | Case | |
|---|---|---|---|---|---|
| System Organ Class Term (SOC) | Preferred Term(PT) | Tri fluvac<br>(N = xx) | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| | | n (%) | n (%) | n (%) | n (%) |
| | | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) | xx(xx.xx) |

**Note**: suspected to be related treatment = probably not related, probably related, definitely related

TREF 2.5: Summary of Adverse Events with Definitely Related and / or Severe

| Study<br>Number | Study<br>Group | Sex | Age | Adverse Event | Start Date | Stop Date | Medication Taken | Severity | Relation | Outcome | *ILI | Serious |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

<sup>\*</sup>ILI-illness like influenza

TREF 2.6: Summary Number of Subjects with Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group

| | Tri fluvac<br>(N = xx) | Comparator<br>(N = xx) |
|---|---|---|
| Illness like Influenza (ILI) | | |
| Yes | | |
| No | | |
| p-value = $xxx$ | | |

Note: This table will be showed number of subjects with and without ILI.

TREF 2.7: Vital Sign of Illness like Influenza (ILI) by GPO Tri fluvac and Active Comparator Group

| | | Tri fluvac<br>(N = xx)* | $\mathbf{(N=xx)^*}$ |
|---|---|---|---|
| Temperature (°C) | | | |
| n | | | |
| Mean(SD) | | | |
| Median | | | |
| Min, Max | | | |
| | P- value = | | |
| Pulse (Beats per m | inute) | | |
| n | | | |
| Mean(SD) | | | |
| Median | | | |
| Min, Max | | | |
| | P- value = | | |
| <b>Blood Pressure</b> | | | |
| Systolic (mmHg) | | | |
| n | | | |
| Mean(SD) | | | |
| Median | | | |
| Min, Max | | | |
| | P- value = | | |
| Diastolic | | | |
| n | | | |
| Mean(SD) | | | |
| Median | | | |
| Min, Max | | | |
| | P- value = | | |

Note: - Vital sign will be compared between GPO Tri fluvac and Active Comparator.

- \* Number of illness like influenza (ILI) events
- Only subject with of illness like influenza (ILI) will be considered for this table.

TREF 2.8: Physical Examination of Illness like Influenza (ILI) Events by GPO Tri fluvac and Active Comparator Group

| | Tri fluvac | Comparator |
|---|---|---|
| | $(\mathbf{N}=\mathbf{x}\mathbf{x})^*$ | $(N = xx)^*$ |
| HEENT, n (%) | | |
| Normal | xx(xx.xx) | xx(xx.xx) |
| Abnormal | xx(xx.xx) | xx(xx.xx) |
| P- value = $x.xxxx$ | | |
| Lungs, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |
| Cardiovascular, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |
| Gastrointestinal, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |
| Musculoskeletal, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |
| Skin, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |
| Neurologic, n (%) | | |
| Normal | | |
| Abnormal | | |
| P- value = | | |

Note: - Physical examination will be compared between GPO Tri fluvac and Active Comparator.

- \* Number of illness like influenza (ILI) events
- Only subject with of illness like influenza (ILI) will be considered for this table.

TREF 2.9: Summary RT- PCR Test for Illness like Influenza (ILI) Events by GPO Tri fluvac and Active Comparator Group

| | Tri fluvac | Comparator |
|---|---|---|
| | $(\mathbf{N}=\mathbf{x}\mathbf{x})^*$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})^*$ |
| Nasal Swab Test Result | | |
| Not done | xx(xx.xx) | xx(xx.xx) |
| Inconclusive | xx(xx.xx) | xx(xx.xx) |
| Influenza A | | |
| Positive | xx(xx.xx) | xx(xx.xx) |
| Negative | xx(xx.xx) | xx(xx.xx) |
| P- value = $x.xxxx$ | | |
| Influenza B | | |
| Positive | xx(xx.xx) | xx(xx.xx) |
| Negative | xx(xx.xx) | xx(xx.xx) |
| P- value = x.xxxx | | |
| Throat Swab Test Result | | |
| Not done | xx(xx.xx) | xx(xx.xx) |
| Inconclusive | xx(xx.xx) | xx(xx.xx) |
| Influenza A | | |
| Positive | xx(xx.xx) | xx(xx.xx) |
| Negative | xx(xx.xx) | xx(xx.xx) |
| P- value = $x.xxxx$ | | |
| Influenza B | | |
| Positive | xx(xx.xx) | xx(xx.xx) |
| Negative | xx(xx.xx) | xx(xx.xx) |
| P- value = x.xxxx | | |
| Conclusion of RT-PCR | | |
| Influenza A H1 | | |
| Influenza A H3 | | |
| Influenza A H5 | | |
| Influenza A unspecified | | |
| Influenza B | | |
| Inconclusive test results | | |
| Influenza not detected | | |
| Other | | |

TREF 2.9: Summary RT-PCR Test for Illness like Influenza (ILI) Events by GPO Tri fluvac and Active Comparator Group (Continue)

| | | Tri fluvac<br>(N = xx)* | Comparator<br>(N = xx)* |
|---|---|---|---|
| Final Diagnosis | | | |
| Influenza | | | |
| ILI | | | |
| Other | | | |
| | P- value = $x.xxxx$ | | |

Note: - Only subject with of illness like influenza (ILI) will be considered for this table.

- \* Number of illness like influenza (ILI) events
- Test result will be compared between GPO Tri fluvac and Active Comparator.

### 3. Post Immunization Reaction

# **Temperature Grading**

- TREF 3.1 Comparison of Temperature Grading at Follow up Visit by GPO Tri Fluvac and Active Comparator Group
- TREF 3.2 Comparison of Temperature Grading at Post Immunization by GPO Tri Fluvac and Active Comparator Group

# Vital Sign

TREF 3.3: Vital Sign by GPO Tri Fluvac and Active Comparator Group

### **Physical Examination**

TREF 3.4: Physical Examination by GPO Tri Fluvac and Active Comparator Group

# Post Immunization Reaction

## **Local Reaction Post Immunization**

- TREF 3.5 Comparison of Maximum Grade of Local Reaction at Post Immunization by GPO

  Tri Fluvac and Active Comparator Group
- TREF 3.6 Comparison of Local Reaction at Post Immunization each Follow up Time by GPO

  Tri Fluvac and Active Comparator Group
- TREF 3.7 Comparison of Maximum Grade of Local Reaction by Symptom at Post Immunization by GPO Tri Fluvac and Active Comparator Group
- TREF 3.8: Summary Number of Local Reaction Days by Symptom at Post Immunization
- TREF 3.9: Summary Number of Local Reaction by Symptom at Post Immunization

## **Systemic Reaction Post Immunization**

- TREF 3.10 Comparison of Maximum Grade of Systemic Reaction at Post Immunization by GPO Tri Fluvac and Active Comparator Group
- TREF 3.11 Comparison of Systemic Reaction at Post Immunization each Follow up Visit by GPO Tri Fluvac and Active Comparator Group
- TREF 3.12 Comparison of Maximum Grade of Systemic Reaction by Symptom at Post Immunization by GPO Tri Fluvac and Active Comparator Group
- TREF 3.13: Summary Number of Systemic Reaction Days by Symptom at Post Immunization
- TREF 3.14: Summary Number of Systemic Reaction by Symptom at Post Immunization

TREF 3.1: Comparison of Temperature Grading at Follow up Visit by GPO Tri Fluvac and Active Comparator Group

| | Tri fluvac | Comparator |
|---|---|---|
| Follow up Visit | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| • | п (%) | n (%) |
| Day 0 | | |
| - Grade 0 | xx(xx.xx) | xx(xx.xx) |
| - Grade 1 | xx(xx.xx) | xx(xx.xx) |
| - Grade 2 | xx(xx.xx) | xx(xx.xx) |
| - Grade 3 | xx(xx.xx) | xx(xx.xx) |
| - Grade 4 | xx(xx.xx) | xx(xx.xx) |
| p - value = x.xxx | X | |
| Day 7 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |
| Day 21 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |
| Day 90 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |

**Note**: Grading of reporting temperature are:

Grade 0: (no) < 38 °C

Grade 1: (mild) 38.0 °C - < 38.6 °C

Grade 2: (moderately high)  $\geq$  38.6 °C - < 39.3 °C

Grade 3: (high)  $\geq 39.3 \, ^{\circ}\text{C} - < 40.0 \, ^{\circ}\text{C}$ 

Grade 4: (Potential Life Threatening) > 40 °C

TREF 3.2: Comparison of Temperature Grading at Post Immunization by GPO Tri Fluvac and Active Comparator Group

| Follow up Visit | Tri fluvac | Comparator |
|---|---|---|
| | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| | n (%) | n (%) |
| 30 min. | | |
| - Grade 0 | xx(xx.xx) | xx(xx.xx) |
| - Grade 1 | xx(xx.xx) | xx(xx.xx) |
| - Grade 2 | xx(xx.xx) | xx(xx.xx) |
| - Grade 3 | xx(xx.xx) | xx(xx.xx) |
| - Grade 4 | xx(xx.xx) | xx(xx.xx) |
| p - value = x.xxxx | | |
| Day 1 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |
| Day 2 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |
| Day 3 | | |
| - Grade 0 | | |
| - Grade 1 | | |
| - Grade 2 | | |
| - Grade 3 | | |
| - Grade 4 | | |
| p - value = | | |

Note: Grading of reporting temperature are:

Grade 0: (no) < 38 °C

Grade 1: (mild) 38.0 °C - < 38.6 °C

Grade 2: (moderately high)  $\geq$  38.6 °C - < 39.3 °C

Grade 3: (high)  $\geq$  39.3 °C -< 40.0 °C

Grade 4: (Potential Life Threatening) > 40 °C

TREF 3.3: Vital Sign at Follow up Visit by GPO Tri Fluvac and Active Comparator Group

| Vital Sign | Da | ay 0 | Da | ay 7 | Da | ny 21 | Da | y 90 |
|---|---|---|---|---|---|---|---|---|
| | Tri fluvac<br>(N = xx) | Comparator $(N = xx)$ | Tri fluvac<br>(N = xx) | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| Temperature (°C) | | | | | | | | |
| n | XX | XX | | | | | | |
| Mean(SD) | xx.xx(xx.xx) | xx.xx(xx.xx) | | | | | | |
| Median | XX.XX | XX.XX | | | | | | |
| Min, Max | XX.XX, XX.XX | XX.XX, XX.XX | | | | | | |
| P- value = | X.X | XXXX | | | | | | |
| Pulse (Beats per | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |
| Min, Max | | | | | | | | |
| P- value = | | | | | | | | |
| <b>Blood Pressure</b> | | | | | | | | |
| Systolic (mmHg) | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |
| Min, Max | | | | | | | | |
| P- value = | | | | | | | | |
| Diastolic | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |

TREF 3.3: Vital Sign at Follow up Visit by GPO Tri Fluvac and Active Comparator Group (Continue)

| Vital Sign | Da | ay 0 | D | ay 7 | Da | ny 21 | Da | y 90 |
|---|---|---|---|---|---|---|---|---|
| | Tri fluvac<br>(N = xx) | Comparator (N = xx) | | Comparator $(N = xx)$ | | Comparator (N = xx) | Tri fluvac<br>(N = xx) | Comparator (N = xx) |
| Min, Max | | | | | | | | |
| P- value = | | | | | | | | |

TREF 3.4: Physical Examination by GPO Tri Fluvac and Active Comparator Group

| | Day 0 | | D | ay 7 | Day 21 | | Day 90 | |
|---|---|---|---|---|---|---|---|---|
| | Tri fluvac | Comparator | Tri fluvac | Comparator | Tri fluvac | Comparator | Tri fluvac | Comparator |
| | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ |
| HEENT, n (%) | | | | | | | | |
| Normal | xx(xx.xx) | xx(xx.xx) | | | | | | |
| Abnormal | xx(xx.xx) | xx(xx.xx) | | | | | | |
| P- value = | X.2 | XXXX | | | | | | |
| Lungs, n (%) | | | | | | | | |
| Normal | | | | | | | | |
| Abnormal | | | | | | | | |
| P- value = | | | | | | | | |
| Cardiovascular, n (%) | | | | | | | | |
| Normal | | | | | | | | |
| Abnormal | | | | | | | | |
| P- value = | | | | | | | | |
| Gastrointestinal, n (%) | | | | | | | | |
| Normal | | | | | | | | |
| Abnormal | | | | | | | | |
| P- value = | | | | | | | | |
| Musculoskeletal, n (%) | | | | | | | | |
| Normal | | | | | | | | |
| Abnormal | | | | | | | | |
| P- value = | | | | | | | | |
| Skin, n (%) | | | | | | | | |
| Normal | | | | | | | | |
| Abnormal | | | | | | | | |
| P- value = | | | | | | | | |

TREF 3.4: Physical Examination by GPO Tri Fluvac and Active Comparator Group (Continue)

| | Da | ay 0 | Da | ay 7 | Da | y 21 | Da | y 90 |
|---|---|---|---|---|---|---|---|---|
| | Tri Fluvac<br>(N = xx) | Comparator (N = xx) | Tri Fluvac<br>(N = xx) | Comparator (N = xx) | Tri Fluvac<br>(N = xx) | - | Tri Fluvac<br>(N = xx) | Comparator (N = xx) |
| Neurologic, n (%) | | | | | | | | |
| Normal | xx(xx.xx) | xx(xx.xx) | | | | | | |
| Abnormal | xx(xx.xx) | xx(xx.xx) | | | | | | |
| P- value = | X.X | XXXX | | | | | | |

TREF 3.5: Comparison of Maximum Grade of Any Local Reaction at Post Immunization by GPO Tri fluvac and Active Comparator Group

| Grade | | Tri Fluvac<br>(N = xx)<br>n (%) | Comparator<br>(N = xx)<br>n (%) |
|---|---|---|---|
| Grade 0 | | xx(xx.xx) | xx(xx.xx) |
| Grade 1 | | xx(xx.xx) | xx(xx.xx) |
| Grade 2 | | xx(xx.xx) | xx(xx.xx) |
| Grade 3 | | xx(xx.xx) | xx(xx.xx) |
| P- value = | X.XXXX | | |

Note: - Any local reaction on any day (by case)

- Erythema and Induration will be not included.

- Grading

Grade 0 - none

Grade 1 - mild

Grade 2 - moderate

Grade 3 - severe

TREF 3.6: Comparison of Local Reaction at Post Immunization each Follow up Time by GPO Tri Fluvac and Active Comparator Group

| | 30 min | | D | ay 1 | D | ay 2 | Da | ay 3 |
|---|---|---|---|---|---|---|---|---|
| Local Reaction | Tri Fluvac<br>(N=xx) | Comparator (N=xx) | Tri Fluvac<br>(N=xx) | Comparator (N=xx) | Tri Fluvac<br>(N=xx) | Comparator (N=xx) | Tri Fluvac<br>(N=xx) | Comparator<br>(N=xx) |
| Pain, n (%) | xx(xx.x) | xx(xx.xx) | | | | | | |
| p-value = | X.2 | xxxx | | | | | | |
| <b>Limitation of arm movement, n (%)</b> p-value = | | | | | | | | |
| - Erythema (cm.) | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |
| Min, Max | | | | | | | | |
| p-value = | | | | | | | | |
| - Swelling (cm.) | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |
| Min, Max | | | | | | | | |
| p-value = | | | | | | | | |
| Induration (cm.) | | | | | | | | |
| n | | | | | | | | |
| Mean(SD) | | | | | | | | |
| Median | | | | | | | | |
| Min, Max | | | | | | | | |
| p-value = | | | | | | | | |

**Note**: - Summary by case who had symptoms

TREF 3.7: Comparison of Maximum Grade of Local Reaction by Symptom at Post Immunization by GPO Tri fluvac and Active Comparator Group

| Local Reaction | | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|---|---|---|---|
| Pain, n (%) | | | |
| Grade 0 | | xx(xx.xx) | xx(xx.xx) |
| Grade 1 | | xx(xx.xx) | xx(xx.xx) |
| Grade 2 | | xx(xx.xx) | xx(xx.xx) |
| Grade 3 | | xx(xx.xx) | xx(xx.xx) |
| p-value = | X.XXXX | | |
| Limitation of arm movemer | ıt, n (%) | | |
| Grade 0 | | | |
| Grade 1 | | | |
| Grade 2 | | | |
| Grade 3 | | | |
| p-value = | | | |

Note: - On any day (by cases)

- Grading

Grade 0 - none Grade 1 - mild Grade 2 - moderate Grade 3 - severe

TREF 3.8: Comparison Number of Subject by Number of Local Reaction Days at Post Immunization GPO Tri fluvac and Active Comparator Group

| Number of Days by Local Reaction | Tri fluvac<br>(N = xx) | $ \begin{array}{c} \text{Comparator} \\ \text{(N = xx)} \end{array} $ |
|---|---|---|
| Pain | | |
| only 30 min. | xx (xx.xx) | xx (xx.xx) |
| 1 day | xx (xx.xx) | xx (xx.xx) |
| 2 days | xx (xx.xx) | xx (xx.xx) |
| 3 days | xx (xx.xx) | xx (xx.xx) |
| p-value = $x.xxxx$ | | |
| Limitation of arm movement | | |
| only 30 min. | xx (xx.xx) | xx (xx.xx) |
| 1 day | xx (xx.xx) | xx (xx.xx) |
| 2 days | xx (xx.xx) | xx (xx.xx) |
| 3 days | xx (xx.xx) | xx (xx.xx) |
| p-value = $x.xxxx$ | | |

Note: - Subjects who had symptom with local reaction will be considered in this table.

- Number of subjects who had symptom will be compared between Tri fluvac and comparator.
- Percentage will be calculated from total enrollment subject.

TREF 3.9: Comparison Number of Subjects by Number of Local Reaction at Post Immunization GPO Tri fluvac and Active Comparator Group

| Number of Local Reaction | Tri fluvac<br>(N = xx) | (N = xx) |
|--------------------------|------------------------|------------|
| No symptom | xx (xx.xx) | xx (xx.xx) |
| 1 symptom | xx (xx.xx) | xx (xx.xx) |
| 2 symptoms | xx (xx.xx) | xx (xx.xx) |
| p-value = $x.xxxx$ | | |

Note: - All enrollment Subjects will be considered in this table.

<sup>-</sup> Percentage will be calculated from total enrollment subject.

TREF 3.10: Comparison of Maximum Grade of Any Systemic Reaction at Post Immunization by GPO Tri fluvac and Active Comparator Group

| Grade | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|---------------------|----------------------|----------------------|
| | n (%) | n (%) |
| Grade 0 | xx(xx.xx) | xx(xx.xx) |
| Grade 1 | xx(xx.xx) | xx(xx.xx) |
| Grade 2 | xx(xx.xx) | xx(xx.xx) |
| Grade 3 | xx(xx.xx) | xx(xx.xx) |
| P- value = $x.xxxx$ | | |

Note: Grading

Grade 0 - none

Grade 1 - mild

Grade 2 - moderate

Grade 3 - severe

TREF 3.11: Comparison of Systemic Reaction at Post Immunization each Follow up Time by GPO Tri fluvac and Active Comparator Group

| | 3 | 0 min | Day 1 Day 2 | | Day 2 | Day 3 | | |
|---|---|---|---|---|---|---|---|---|
| Systemic Reaction | Tri<br>fluvac | Comparator<br>(N=xx) | Tri fluvac<br>(N=xx) | Comparator (N=xx) | Tri fluvac<br>(N=xx) | Comparator (N=xx) | Tri fluvac<br>(N=xx) | Comparator (N=xx) |
| - <b>Headache, n (%)</b><br>p-value = | XX(XX.XX) | XX(XX.XX) | | | | | | |
| - <b>Fatigue, n (%)</b><br>p-value = | | | | | | | | |
| - <b>Malaise, n (%)</b><br>p-value = | | | | | | | | |
| - Chills, n (%)<br>p-value = | | | | | | | | |
| - <b>Myalgia, n (%)</b><br>p-value = | | | | | | | | |
| - <b>Arthralgia, n (%)</b><br>p-value = | | | | | | | | |
| - <b>Nausea, n (%)</b><br>p-value = | | | | | | | | |
| - <b>Vomiting, n (%)</b><br>p-value = | | | | | | | | |
| - <b>Rash, n (%)</b><br>p-value = | | | | | | | | |

Note: Summary by case who had symptoms

TREF 3.12: Comparison of Maximum Grade of Systemic Reaction by Symptom at Post Immunization by GPO Tri fluvac and Active Comparator Group

| Systemic Reaction | Tri fluvac<br>(N=xx) | Comparator (N=xx) |
|-------------------|----------------------|-------------------|
| Headache, n (%) | , , | ` ' |
| Grade 0 | xx(xx.xx) | xx(xx.xx) |
| Grade 1 | XX(XX.XX) | xx(xx.xx) |
| Grade 2 | xx(xx.xx) | xx(xx.xx) |
| Grade 3 | xx(xx.xx) | xx(xx.xx) |
| p-value = x.xxxx | | |
| Fatigue, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |
| Malaise, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |
| Chills, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |
| Myalgia, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |
| Arthralgia, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |

TREF 3.12: Comparison of Maximum Grade of Systemic Reaction by Symptom at Post Immunization by GPO Tri fluvac and Active Comparator Group (Continue)

| Systemic Reaction | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|-------------------|----------------------|----------------------|
| Nausea, n (%) | | |
| Grade 0 | xx(xx.xx) | xx(xx.xx) |
| Grade 1 | xx(xx.xx) | xx(xx.xx) |
| Grade 2 | XX(XX.XX) | xx(xx.xx) |
| Grade 3 | xx(xx.xx) | xx(xx.xx) |
| p-value = | | |
| Vomiting, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |
| Rash, n (%) | | |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| p-value = | | |

Note: • On any day (by cases)

Grading

Grade 0 - none

Grade 1 - mild

Grade 2 - moderate

Grade 3 - severe

TREF 3.13: Comparison Number of Subject by Number of Systemic Reaction Days at Post Immunization GPO Tri fluvac and Active Comparator Group

| Number ( | of Days by Systemic Reaction | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|---|---|---|---|
| Headache | only 30 min. | xx(xx.xx) | xx(xx.xx) |
| | 1 day | xx(xx.xx) | xx(xx.xx) |
| | 2 days | xx(xx.xx) | xx(xx.xx) |
| | 3 days | xx(xx.xx) | xx(xx.xx) |
| | 4 days | xx(xx.xx) | xx(xx.xx) |
| | 5 days | xx(xx.xx) | xx(xx.xx) |
| | p-value = $x.xxxx$ | | |
| Fatigue | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |
| Malaise | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |
| Chills | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |
| Myalgia | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |

TREF 3.13: Comparison Number of Subject by Number of Systemic Reaction Days at Post Immunization between GPO Tri fluvac and Active Comparator Group (Continue)

| Number of Days by Systemic Reaction | | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|---|---|---|---|
| Arthralgia | only 30 min. | XX(XX.XX) | XX(XX.XX) |
| | 1 day | xx(xx.xx) | xx(xx.xx) |
| | 2 days | xx(xx.xx) | xx(xx.xx) |
| | 3 days | xx(xx.xx) | xx(xx.xx) |
| | 4 days | xx(xx.xx) | xx(xx.xx) |
| | 5 days | xx(xx.xx) | xx(xx.xx) |
| | p-value = $x.xxxx$ | | |
| Nausea | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |
| Vomiting | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |
| Rash | only 30 min. | | |
| | 1 day | | |
| | 2 days | | |
| | 3 days | | |
| | 4 days | | |
| | 5 days | | |
| | p-value = $x.xxxx$ | | |

Note: - Subjects who had symptom with Systemic reaction will be considered in this table.

- Number of subjects who had symptom will be compared between Tri fluvac and comparator.
- Percentage will be calculated from total enrollment subjects.

TREF 3.14: Comparison Number of Subjects by Number of Systemic Reaction at Post Immunization between GPO Tri fluvac and Active Comparator Group

| Number of Local Reaction | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
|--------------------------|----------------------|----------------------|
| No symptom | xx(xx.xx) | XX(XX.XX) |
| 1 symptom | xx(xx.xx) | xx(xx.xx) |
| 2 symptoms | xx(xx.xx) | xx(xx.xx) |
| 3 symptoms | xx(xx.xx) | xx(xx.xx) |
| 4 symptoms | xx(xx.xx) | xx(xx.xx) |
| 5 symptoms | xx(xx.xx) | xx(xx.xx) |
| 6 symptoms | xx(xx.xx) | xx(xx.xx) |
| 7 symptoms | xx(xx.xx) | xx(xx.xx) |
| 8 symptoms | xx(xx.xx) | xx(xx.xx) |
| 9 symptoms | xx(xx.xx) | xx(xx.xx) |

Note: - All enrollment Subjects will be considered in this table.

<sup>-</sup> Percentage will be calculated from total enrollment subject.

# 4. Immunogenicity

- TREF 4.1: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90
- TREF 4.2: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator at Any Day
- TREF 4.3: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer < 1:10
- TREF 4.4: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer ≥ 1:10
- TREF 4.5: Comparing Seroprotective Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90
- TREF 4.6: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer < 1:10
- TREF 4.7: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer  $\geq 1:10$
- TREF 4.8: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group
- TREF 4.9: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer < 1:10
- TREF 4.10: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer  $\geq 1:10$
- TREF 4.11: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group
- TREF 4.12: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer < 1:10
- TREF 4.13: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer ≥ 1:10

TREF 4.1: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90

| HI Assay | Follow up Day | Study Group | 4- fold rising<br>n (%) | Not 4 -fold<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | X | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu A H3 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxxx | | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu B | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | x | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |

Note: Enrollment cases will be compared between GPO Tri fluvac and Active Comparator Group.
TREF 4.2: Comparing Seroconversion Rates between GPO Tri fluvac and Active Comparator at Any Day

| HAI Assay | Study Group | 4- fold rising<br>n (%) | Not 4 -fold<br>n (%) |
|---|---|---|---|
| H1 Antibody Titer | Tri fluvac $(N = xx)$<br>Comparator $(N = xx)$<br>p - value = x.xxxx | xx.xx(xx.xx)<br>xx.xx(xx.xx) | xx.xx(xx.xx)<br>xx.xx(xx.xx) |
| H3 Antibody Titer | Tri fluvac $(N = xx)$<br>Comparator $(N = xx)$<br>p - value = | | |
| Flu B Antibody Titer | Tri fluvac $(N = xx)$<br>Comparator $(N = xx)$<br>p - value = | | |

TREF 4.3: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub - Group Pre-Vaccination HI Antibody titer < 1:10

| HI Assay | Follow up Day | Study Group | 4- fold rising<br>n (%) | Not 4 -fold<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = $x$ | .XXXX | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = $x$ | .XXXX | |
| Flu A H3 | Day 21 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu B | Day 21 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| | <b>Day 90</b> | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |

TREF 4.4: Comparing Seroconversion Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer  $\geq 1:10$ 

| HI Assay | Follow up Day | Study Group | 4- fold rising<br>n (%) | Not 4 -fold<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=x | x) xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx | x) xx(xx.xx) | xx(xx.xx) |
| | | p - va | lue = x.xxxx | |
| | <b>Day 90</b> | Tri fluvac (N=x | x) | |
| | | Comparator (N=xx | <b>x</b> ) | |
| | | p - va | lue = | |
| Flu A H3 | Day 21 | Tri fluvac (N=x | x) xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx | x $xx(xx.xx)$ | xx(xx.xx) |
| | | p - va | lue = x.xxxx | |
| | <b>Day 90</b> | Tri fluvac (N=x | x) | |
| | | Comparator (N=xx | x) | |
| | | p - va | lue = | |
| Flu B | Day 21 | Tri fluvac (N=x | x) xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx | x) xx(xx.xx) | xx(xx.xx) |
| | | p - va | lue = x.xxxx | |
| | <b>Day 90</b> | Tri fluvac (N=x | x) | |
| | | Comparator (N=xx | x) | |
| | | p - va | lue = | |

TREF 4.5: Comparing Seroprotective Rates between GPO Tri fluvac and Active Comparator Group Separated by HI Assay at Day 21 and 90

| HI Assay | Follow up Day | Study Group | Seroprotective<br>n (%) | Non-seroprotective<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxxx | | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu A H3 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxxx | | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu B | <b>Day 21</b> | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxxx | | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |

<sup>-</sup> Seroprotective level: HI antibody titer  $\geq 1:40$ 

TREF 4.6: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer < 1:10

| HI Assay | Follow up Day | Study Group | Seroprotective<br>n (%) | Non-seroprotective<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | XX | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu A H3 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | XX | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu B | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | xx | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |

TREF 4.7: Comparing Seroprotective Rates Separated by HI Assay at Day 21 and 90 in Sub-Group Pre-Vaccination HI Antibody titer ≥ 1:10

| HI Assay | Follow up Day | Study Group | Seroprotective<br>n (%) | Non-seroprotective<br>n (%) |
|---|---|---|---|---|
| Flu A H1 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | XX | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu A H3 | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | XX | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |
| Flu B | Day 21 | Tri fluvac (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | Comparator (N=xx) | xx(xx.xx) | xx(xx.xx) |
| | | p - value = x.xxx | xx | |
| | Day 90 | Tri fluvac (N=xx) | | |
| | | Comparator (N=xx) | | |
| | | p - value = | | |

TREF 4.8: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group

| HAI Assay | Day 0<br>GMT(95% CI) | Day 21<br>GMT(95% CI) | Day 90<br>GMT(95% CI) |
|---|---|---|---|
| Flu A H1 Antibody titer | | | |
| Tri fluvac | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Comparator | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| P - value = | X.XXXX | X.XXXX | X.XXXX |
| Flu A H3 Antibody titer | | | |
| Tri fluvac | | | |
| Comparator | | | |
| P - value = | | | |
| Flu B Antibody titer | | | |
| Tri fluvac | | | |
| Comparator | | | |
| P - value = | | | |

TREF 4.9: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer < 1:10

| HAI Assay | Day 0<br>GMT(95% CI) | Day 21<br>GMT(95% CI) | Day 90<br>GMT(95% CI) |
|---|---|---|---|
| Flu A H1 Antibody titer | | | |
| Tri fluvac | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Comparator | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| P - value = | X.XXXX | X.XXXX | X.XXXX |
| Flu A H3 Antibody titer | | | |
| Tri fluvac | | | |
| Comparator | | | |
| P - value = | | | |
| Flu B Antibody titer | | | |
| Tri fluvac | | | |
| Comparator | | | |
| P - value = | | | |

- † For titer reported as < 10, a value of 5 will be assigned when computing GMT

TREF 4.10: Geometric Mean Titer (GMTs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer ≥ 1:10

| HAI A | ssay | Day 0<br>GMT(95% CI) | Day 21<br>GMT(95% CI) | Day 90<br>GMT(95% CI) |
|---|---|---|---|---|
| Flu A H1 Ant | tibody titer | | | |
| Tri fluvac | | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Comparator | | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| | P - value = | x.xxxx | X.XXXX | x.xxx |

## Flu A H3 Antibody titer

Tri fluvac

Comparator

P - value =

### Flu B Antibody titer

Tri fluvac

Comparator

P - value =

Note: - Enrollment cases will be compared between GPO Tri fluvac and Active Comparator.

-  $\dagger$  For titer reported as < 10, a value of 5 will be assigned when computing GMT

TREF 4.11: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group

| II A I A seev | Tri fluvac | Comparator |
|---|---|---|
| HAI Assay | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| Flu A H1 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Day 21 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | xx.xx | XX.XX |
| Day 90 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | XX.XX | XX.XX |
| Flu A H3 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| GMFRs <sup>‡</sup> | | |
| Day 90 | | |
| GMT † (95% CI) | | |
| GMFRs <sup>‡</sup> | | |
| Flu B antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| $\mathrm{GMFRs}^{\ddagger}$ | | |
| <b>Day 90</b> | | |
| GMT <sup>†</sup> (95% CI) | | |
| GMFRs <sup>‡</sup> | | |

-  $\dagger$  For titer reported as < 10, a value of 5 will be assigned when computing GMT;  $\ddagger$  GMFR is the geometric mean of the ratios of post - vaccination to the pre-vaccination

TREF 4.12: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer < 1:10

| II A I A seev | Tri fluvac | Comparator |
|---|---|---|
| HAI Assay | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| Flu A H1 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Day 21 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | xx.xx | XX.XX |
| Day 90 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | XX.XX | XX.XX |
| Flu A H3 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| GMFRs <sup>‡</sup> | | |
| Day 90 | | |
| GMT † (95% CI) | | |
| GMFRs <sup>‡</sup> | | |
| Flu B antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| $\mathrm{GMFRs}^{\ddagger}$ | | |
| <b>Day 90</b> | | |
| GMT <sup>†</sup> (95% CI) | | |
| GMFRs <sup>‡</sup> | | |

-  $\dagger$  For titer reported as < 10, a value of 5 will be assigned when computing GMT;  $\ddagger$  GMFR is the geometric mean of the ratios of post - vaccination to the pre-vaccination

TREF 4.13: Geometric Mean Fold Rises (GMFRs) of Immune Response by GPO Tri fluvac and Active Comparator Group in Sub-Group Pre-Vaccination HI Antibody Titer ≥ 1:10

| TIAL Assess | Tri fluvac | Comparator |
|---|---|---|
| HAI Assay | $(\mathbf{N} = \mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| Flu A H1 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| Day 21 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | xx.xx | XX.XX |
| Day 90 | | |
| $GMT^{\dagger}$ (95% CI) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| GMFRs | xx.xx | XX.XX |
| Flu A H3 antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| $\mathrm{GMFRs}^{\ddagger}$ | | |
| Day 90 | | |
| GMT † (95% CI) | | |
| $\mathrm{GMFRs}^{\ddagger}$ | | |
| Flu B antibody titer | | |
| Day 0 | | |
| GMT † (95% CI) | | |
| Day 21 | | |
| GMT † (95% CI) | | |
| $\mathrm{GMFRs}^{\ddagger}$ | | |
| <b>Day 90</b> | | |
| GMT † (95% CI) | | |
| GMFRs <sup>‡</sup> | | |

-  $\dagger$  For titer reported as < 10, a value of 5 will be assigned when computing GMT;  $\ddagger$  GMFR is the geometric mean of the ratios of post - vaccination to the pre-vaccination

### 5. Concomitant Medication

TREF 5: Summary of Concomitant Medication According to WHO DD by GPO Tri fluvac and Active Comparator Group

TREF 5: Summary of Concomitant Medication According to WHO DD by GPO Tri fluvac and Active Comparator Group

| | | Number | of Event | Number of Case | |
|---|---|---|---|---|---|
| Anatomical Main Group | Therapeutic Subgroup | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) | Tri fluvac<br>(N=xx) | Comparator<br>(N=xx) |
| | | n (%) | n (%) | n (%) | n (%) |
| xxxxxxxx | xxxxxxxx | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| XXXXXXXX | xxxxxxxx | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

#### APPENDICES

Appendix 01: Listing of Subjects were Excluded from Analysis

| Observe | Screening Number | Reason for Exclude |
|---------|------------------|--------------------|
| 1 | | |
| 2 | | |
| 3 | | |
| ••• | | |

Appendix 02: Listing of Past Medical History and Pre-existing Condition in Last 6 Months

| Observe Subject<br>Number | Study<br>Group | Diagnosis<br>/Symptoms<br>/Signs | Month/Year started | Currently active? |
|---|---|---|---|---|
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

# Appendix 03: Listing of Past Immunization History in Last 6 Months

| Observe Subject<br>Number | Study<br>Group | Immunization | Month/Year started | Completed? |
|---|---|---|---|---|
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

Appendix 04: Listing of Local Reaction at Post Immunization

| | Subject | | | |
|---------|---------|-------------|---------|-----------------------|
| Observe | Number | Study Group | Symptom | Follow up Day (Grade) |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

# Appendix 05: Listing of Systemic Reaction at Post Immunization

| Observe | Subject Number | Study Group | Symptom | Follow up Day (Grade) |
|---------|----------------|-------------|---------|-----------------------|
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |

## Appendix 06: Listing of Adverse Event

3

| No. | Subject<br>Number | Seq. | Adverse<br>Event | Start<br>Date | End<br>Date | AEs (hrs) | Medication<br>taken? | Severity | Related<br>to<br>Study<br>Vac | Outcome | AE-<br>Serious<br>? | Date of<br>Immunization | Study<br>Group | #Day at AE<br>started after<br>Immunization |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | | | | | | | | | | | | | _ |
| 2 | | | | | | | | | | | | | | |

Note: #Day at AE started after immunization date will be calculated from date of immunization to date at AE started.

## Appendix 07: Listing of Illness like Influenza (ILI)

| | • • • | | | | ` | , | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | Subject<br>Number | ILI<br>Seq. | Specimen<br>Collection<br>Date | Date of<br>Receipt | Time of<br>Receipt | Nasal swab<br>Test | Result | Nasal swab<br>Result<br>Influenza B | Throat Swab<br>Test | Result | Throat<br>swab<br>Result<br>Influenza<br>B | Conclusion<br>of RT-PCR | Final<br>Diagnosis |
| 1 | | | | | | | | | | | | | |
| 2 | | | | | | | | | | | | | |
| 3 | | | | | | | | | | | | | |
| | Note: | | | | | | | | | | | | |

## **Appendix 08: Listing of Concomitant Medication**

| No | Subject<br>Number | Study Group | Dose | Unit | Route Frequency | Start<br>Date | End date | Ongoing | Indication | Date of<br>Immunization | #Day of<br>Conmed<br>started after<br>Immunization |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | | | | | | | | | | |
| 2 | | | | | | | | | | | |
| 3 | | | | | | | | | | | |

Note: #Day at Conmed started after immunization will be calculated from date of immunization to date of Conmed started.

Appendix 09: List of HAI Assay (Flu A H1 Antigen)

| Study number | Day 0 | Day 21 | Day 90 | Study Group |
|--------------|-------|--------|--------|-------------|
| 1 | XX | XX | XX | XX |
| 2 | XX | XX | XX | XX |
| 3 | | | | |
| ••• | | ••• | ••• | ••• |

**Note**: For titer reported as < 10, a value of 5 will be assigned.

Appendix 10: List of HAI Assay (Flu A H3 Antigen)

| Study number | Day 0 | <b>Day 21</b> | Day 90 | Study Group |
|--------------|-------|---------------|--------|-------------|
| 1 | XX | XX | XX | XX |
| 2 | XX | XX | XX | XX |
| 3 | | | | |
| ••• | | ••• | | |

**Note**: For titer reported as < 10, a value of 5 will be assigned.

Appendix 11: List of HAI Assay (Flu B Antigen)

| Study number | Day 0 | Day 21 | Day 90 | Study Group |
|--------------|-------|--------|--------|-------------|
| 1 | XX | XX | XX | XX |
| 2 | XX | XX | XX | XX |
| 3 | | | | |
| ••• | | ••• | ••• | ••• |

**Note**: For titer reported as < 10, a value of 5 will be assigned.